CLINICAL TRIAL: NCT06615960
Title: The Safety and Effectiveness of PANAF- Premium TM Snake Venom Antiserum-Pan Africa Administered As a Standard Treatment for Cases of Snakebites- a Phase IV Open Label Trial
Brief Title: Safety and Effectiveness of PANAF-Premium TM Snake Venom Antiserum As Standard Treatment for Snakebites
Acronym: PMS
Status: Recruiting | Type: Observational
Sponsor: Premium Serums & Vaccines Pvt.Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PMS1001
Record Dates: First submitted 2024-09-08; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Snake Bites
MeSH Terms: conditions — Snake Bites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Snakebite envenomation (SBE) is a major public health problem in many developing countries. Standard snake antivenom (SA) remains the primary treatment and has been shown to reduce mortality in observational studies conducted in several sub-Saharan African (SSA) countries. Although it is relatively available in other endemic contexts such as Asia and Latin America, there have been major challenges with the reliable supply of effective products in sub-Saharan Africa for many years. Premium Serums & Vaccines Pvt. Ltd. (PSVPL) recently introduced its SA brand, namely PANAF-Premium TM, manufactured to address unmet treatment needs in the local context. This serum has received WHO approval for use in sub-Saharan Africa and is used in Cameroon with neutralizing efficacy for 24 species represented in Africa.

This is an open-label, Phase IV post-marketing surveillance study to collect safety and effectiveness data systematically following the administration of PANAF-Premium TM. The study will describe the types, severity, and number of adverse events recorded following the administration of PANAF-Premium TM and its effectiveness for snakebite management. Epidemiological data will also be collected, along with information on the snake species typically responsible for bites in the North region of Cameroon, the type of envenomation, the total dose of SA required for reversal of envenomation, and the total time required for clinical recovery. This will complement the international and national pool of pharmacovigilance data.

DETAILED DESCRIPTION:
Background: Snakebite envenomation (SBE) is a major public health problem in many developing countries. Conventional snake antivenom (SA) remains the primary treatment and has been shown to reduce mortality in observational studies conducted in several sub-Saharan African (SSA) countries. Although it is relatively available in other endemic contexts such as Asia and Latin America, there have been major challenges with the reliable supply of effective products in sub-Saharan Africa for many years. Premium Serums & Vaccines Pvt. Ltd. (PSVPL) recently introduced its SA brand, namely PANAF-Premium TM, manufactured to the latest standards, providing a solution to address unmet treatment needs in the local context. This serum has received WHO approval for use in sub-Saharan Africa and is used in Cameroon with neutralizing efficacy for 24 species represented in Africa. Since antivenom is of animal origin, it can cause adverse reactions ranging from mild itching to fatal anaphylaxis; therefore, patients should be treated appropriately or given prophylactic premedication. Approximately 20% of cases may develop early (within a few hours) or late (five days or more) allergic reactions after administration of snake antivenom. This open-label, Phase IV post-marketing surveillance study aims to collect safety and effectiveness data systematically following administration of PANAF-Premium TM. The study will describe the types, severity, and number of adverse events recorded following administration of PANAF-Premium TM and its effectiveness for snakebite management. Additionally, epidemiological data will be collected regarding the snake species typically responsible for bites in the North Cameroon region, the type of envenomation, the total dose of SA required for reversal of envenomation, and the total time required for clinical recovery. This will also contribute to the international and national pool of pharmacovigilance data.

Method: An open-label, Phase IV post-marketing surveillance trial will be conducted to describe the types, severity, and number of adverse events recorded during snakebite management. The average dose of SA used will be identified, and the duration of recovery, as well as the type of snakes prevalent in the area, will be explored. Eligible patients will be admitted to the hospital, and case management will be in accordance with the standard protocol followed in Cameroon and adapted from the guidelines of the African Society of Venomology. Any medication or procedure necessary to save the patient will be permitted. If antivenom serum is needed, the study drug to be used is PANAF-Premium TM (Snake Venom Antiserum-Pan Africa), manufactured by Premium Serums & Vaccines Pvt. Ltd. Any suspicious or unexpected serious adverse events (SAEs) will be recorded immediately and reported to the sponsor/ethics committee for further action. There will be no restrictions on the use of any concomitant medication or other interventions or investigations mandated by the patient's clinical condition.

ELIGIBILITY:
Inclusion Criteria:

Patients of both sex and of any age, with history of snakebites/unknown bites received in study sites

* Willingness to participate in the study by signing the Informed Consent Form (ICF)
* Presence of one or more signs of envenomation detected by clinical examination including positive clot test. Patient may present with one or more of following visible clinical signs and symptoms of snake envenomation being local or systemic -

Defining local and systemic envenomation

1. Local envenomation- (I) Presence of bite marks with or without oozing of blood, blistering and change in color of skin.

   (ii) Rapidly progressive or massive swelling involving more than half of the bitten limb within few hours of bite (without tourniquet) (iii) Development of enlarged tender lymph nodes draining the bitten part within couple of hours after bite
2. Systemic envenomation- (i) Neurotoxic syndrome- signs of neuro-paralysis like blurring of vision, double vision, difficulty in swallowing, sleepy feeling, drooping of head, slurring of speech and the voice may become indistinct with shallow breathing, ptosis, ataxia, respiratory paralysis and generalized flaccid paralysis.

(ii) Hemotoxic syndrome- spontaneous systemic bleeding, nausea, vomiting, abdominal pain and abdominal tenderness suggestive of gastro-intestinal or retro-peritoneal bleed and/or renal damage, coagulopathy detected by 20 min WBCT with or without external bleeding and shock and a clinical condition/envenomation serious enough to administer SA will be eligible for enrolment

Exclusion Criteria:

* Participants not able to give consent
* Participants who are unable to understand the nature, scope, significance and consequences of this clinical trial
* Pre-existing renal disease, uncontrolled chronic obstructive airway disease, congestive heart failure or previous myocardial infarction and consumption of diuretics, anticoagulants and antiplatelet drugs have been causes for exclusion in a few earlier studies as these illnesses and medications could have altered the clinical and laboratory profile of patients with envenomation.
* Known history of hypersensitivity to the investigational drug or to drugs with a similar chemical structure
* Simultaneous participation in any clinical trial involving administration of an investigational medicinal product within 30 days prior to clinical trial beginning
* Participants with a physical or psychiatric condition which at the investigator's discretion may put the subject at risk, may confound the trial results, or may interfere with the subject's participation in this clinical trial
* Known or persistent abuse of medication, drugs or alcohol Others conditions may include evidence of clinically significant neurological, cardiac, pulmonary, hepatic or renal disease as far as can be assessed by history of participants, physical examination, and/or laboratory examinations.

NB: Patient previously sensitized with equine antiserum such as Tetanus or Diphtheria antitoxin or patients having received treatment with adrenaline, antihistamine, or steroids as a part of treatment at primary health care center and pregnancy will not be excluded. Since this is a post-marketing study, these patients will be included, and this information will be factored in while collating and analyzing data.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit participants with a history of snakebites or unknown bites showing signs of envenomation requiring Snake Antiserum. Participants will come from health districts in Mayo Oulo, Gashiga, Poli, and Garoua I, located in the North region of Cameroon. One facility in each district has been selected based on prior snakebite cases: Garoua Regional Hospital, Poli District Hospital, Mayo Oulo District Hospital, and Gashiga District Hospital. No specific gender ratio is required, as previous studies have shown no differences in treatment effectiveness or safety between genders.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-02-26 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Safety of Panaf Premuim | 30 days
  Measured by the frequency and severity of the recorded Adverse events based on clinical evaluation using DAAD (Division of AIDS grading of AE) grading classification.
Safety of Panaf Premium | 30 days
  Measured by the factors associated with the occurrence of adverse events, assessed through clinical evaluation and review of concomitant medication.
Effectiveness of Panaf Premium | 30 days
  Measured by the number of days required to control toxicity, defined as the time in days to achieve reversal of a positive Whole Blood Clotting Test (WBCT) in cases of hemotoxic envenomation, and/or the time to reverse clinical signs and symptoms based on the African Society of Venimology's classification and grading of envenomation.
Effectiveness of Panaf Premium | 30 days
  Effectiveness will be measured by the average dose of snake antivenom administered and documented throughout the patient's follow-up, with complete recovery defined by the resolution of symptoms according to the African Society of Venimology's classification and grading system

SECONDARY OUTCOMES:
Identification of Snake Species Responsible for Envenomation | 6 months
  This outcome will be assessed by identifying the snake species responsible for envenomation, based on the description provided by the patient, clinical evaluation, and, where available or laboratory analysis. The investigator will document the snake species involved using classification systems as per guidelines of the African Society of Venimology
Snake bite epidemiology | 6 months
  This outcome will be assessed by calculating the proportion of patients who present with envenomation, categorized by age, sex, and clinical syndrome (e.g., neurotoxic, hemotoxic, or cytotoxic). Data will be collected using patient demographic information, clinical assessments, and envenomation classification systems based on the African Society of Venimology guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Khadillar, Study Director — Premuim serums
Locations (1):
- Garoua Regional Hospital, Garoua, North Region, Cameroon

IPD SHARING:
Plan to Share IPD: Undecided
This has not yet been decided for the moment

REFERENCES:
- [Background] Gutierrez JM, Calvete JJ, Habib AG, Harrison RA, Williams DJ, Warrell DA. Snakebite envenoming. Nat Rev Dis Primers. 2017 Sep 14;3:17063. doi: 10.1038/nrdp.2017.63. PMID 28905944
- [Background] Visser LE, Kyei-Faried S, Belcher DW. Protocol and monitoring to improve snake bite outcomes in rural Ghana. Trans R Soc Trop Med Hyg. 2004 May;98(5):278-83. doi: 10.1016/S0035-9203(03)00065-8. PMID 15109550
- [Background] Schiermeier Q. Africa braced for snakebite crisis. Nature. 2015 Sep 17;525(7569):299. doi: 10.1038/525299a. No abstract available. PMID 26381961
- [Background] Chippaux JP, Habib AG. Antivenom shortage is not circumstantial but structural. Trans R Soc Trop Med Hyg. 2015 Dec;109(12):747-8. doi: 10.1093/trstmh/trv088. No abstract available. PMID 26626337
- [Background] Brown NI. Consequences of neglect: analysis of the sub-Saharan African snake antivenom market and the global context. PLoS Negl Trop Dis. 2012;6(6):e1670. doi: 10.1371/journal.pntd.0001670. Epub 2012 Jun 5. PMID 22679521
- [Background] Gutierrez JM. Global Availability of Antivenoms: The Relevance of Public Manufacturing Laboratories. Toxins (Basel). 2018 Dec 24;11(1):5. doi: 10.3390/toxins11010005. PMID 30586868
- [Background] Potet J, Smith J, McIver L. Reviewing evidence of the clinical effectiveness of commercially available antivenoms in sub-Saharan Africa identifies the need for a multi-centre, multi-antivenom clinical trial. PLoS Negl Trop Dis. 2019 Jun 24;13(6):e0007551. doi: 10.1371/journal.pntd.0007551. eCollection 2019 Jun. PMID 31233536
- [Background] Habib AG, Warrell DA. Antivenom therapy of carpet viper (Echis ocellatus) envenoming: effectiveness and strategies for delivery in West Africa. Toxicon. 2013 Jul;69:82-9. doi: 10.1016/j.toxicon.2013.01.002. Epub 2013 Jan 20. PMID 23339853